CLINICAL TRIAL: NCT03159260
Title: The Effect of Theraworx/[pH]Uel on Night-time Leg Cramps and Spasm Symptoms Including Quality of Life, Depression and Sleep Quality
Brief Title: Effect of Theraworx/[pH]Uel on Night-time Leg Cramps and Spasm Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LegCramp
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Leg Cramp, Nocturnal
Keywords: night-time leg cramps; topical; spasm
MeSH Terms: conditions — Sleep-Wake Transition Disorders; Spasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Product has come in identical bottles from manufacturer. Both the investigators and statistician will remind blind until the conclusion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Theraworx (Experimental): Subjects will receive two 3 ounce foam dispensers corresponding to their group assignment (Foam A or Foam B) and a 2-week Compliance and Symptom Log. The contents of these two foams will remain blind to the subjects and the data collectors until all 50 subjects complete the study protocol. One of the foams will contain Theraworx/[pH]uel (treatment) and the other will contain a physiologically inert substance (placebo control).
  Interventions: Device: Theraworx
- Placebo (Placebo Comparator): Subjects will receive two 3 ounce foam dispensers corresponding to their group assignment (Foam A or Foam B) and a 2-week Compliance and Symptom Log. The contents of these two foams will remain blind to the subjects and the data collectors until all 50 subjects complete the study protocol. One of the foams will contain Theraworx/[pH]uel (treatment) and the other will contain a physiologically inert substance (placebo control).
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Theraworx — Subjects will be instructed to apply the topical foam they have been assigned to their entire upper and lower legs and feet using 8 pumps from the product dispenser per leg (upper thigh to foot) before retiring each evening for the next 14 days. If subjects experience leg cramps or spasms after retiring they will be instructed to reapply to 2 pumps of the foam to the affected area in response to each event. Each morning during the 14 days in which subjects apply the foam they will be asked to complete the Compliance and Symptom Log that documents the incidence and severity of night-time cramps and spasms their use of the foam and any other therapies they used to treat their night-time cramps and spasm.
  Arms: Theraworx
Other: Placebo — Subjects will be instructed to apply the topical foam they have been assigned to their entire upper and lower legs and feet using 8 pumps from the product dispenser per leg (upper thigh to foot) before retiring each evening for the next 14 days. If subjects experience leg cramps or spasms after retiring they will be instructed to reapply to 2 pumps of the foam to the affected area in response to each event. Each morning during the 14 days in which subjects apply the foam they will be asked to complete the Compliance and Symptom Log that documents the incidence and severity of night-time cramps and spasms their use of the foam and any other therapies they used to treat their night-time cramps and spasm.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of Theraworx/[pH]uel on the frequency and severity of night-time cramps and spasms symptoms, including quality of life, depression and sleep quality when compared to a placebo.

DETAILED DESCRIPTION:
50 subjects who claim to have experienced night-time cramps and spasms on average at least three times per week will be recruited. Eligible individuals will be scheduled to attend a "consent and baseline assessment" (T1). During this visit, the study will be described by a member of the research team and the subjects will be asked to provide written consent to participate in the protocol. Following providing informed consent, the subjects will be asked to complete a series of questionnaires about their demographic characteristics, presence and severity of night-time cramps and spasms symptoms, including quality of life, depression and sleep quality. Once these questionnaires are completed all subjects will complete a 14-day no treatment period in which they will be told to engage in their usual activities and treatments. Subjects will return following this two week period (T2) and complete the same questionnaires. Variables that will be collected at T2 include presence and severity of night-time cramps and spasm symptoms, including quality of life, depression and sleep quality. Subjects will be asked to refer their responses on these instruments to the previous 2 weeks following completion of the baseline assessment. Once the subjects have completed these instruments they will be randomly assigned to one of two study groups with 25 of in "Foam A" and 25 in"Foam B." Subjects will receive two 3 ounce foam dispensers corresponding to their group assignment (Foam A or Foam B) and a 2-week Compliance and Symptom Log. Subjects will be instructed to apply the topical foam they have been assigned to their entire upper and lower legs and feet using 8 pumps from the product dispenser per leg (upper thigh to foot) before retiring each evening for the next 14 days. If subjects experience leg cramps or spasms after retiring they will be instructed to reapply to 2 pumps of the foam to the affected area in response to each event. Each morning during the 14 days in which subjects apply the foam they will be asked to complete the Compliance and Symptom Log that documents the incidence and severity of night-time cramps and spasms their use of the foam and any other therapies they used to treat their night-time cramps and spasm. Following 14 consecutive days of applying the assigned foam, subjects will return to SSR (T3) and return the completed Treatment Compliance Log to the research staff. During this final visit subjects will again complete the same questionnaires that were completed during the T2 visit, referring the responses to the previous 2 weeks when the subjects were applying the assigned foam to the legs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who claim to have experienced night-time cramps and spasms on average at least three times per week

Exclusion Criteria:

* Individuals will be excluded from the study if they are pregnant, have been previously diagnosed with a non-RLS sleep disorder, previously diagnosed with schizophrenia or any other neurological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Spine Rehab, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Theraworx: Participants received 2, 3 ounce foam dispensers corresponding to their group (FoamA or FoamB) and a 2-week Compliance and Symptom Log. The participants were blind to the contents of the foam and the investigators until the study was completed. One foam contained Theraworx/[pH]uel (treatment) and the other contained a physiologically inert substance (placebo control).
  Theraworx: Participants were instructed to apply the assigned foam to their entire upper and lower legs and feet using 8 pumps from the dispenser per leg before retiring each evening for 14 days. If participants experienced leg cramps or spasms after retiring they were instructed to reapply 2 pumps of the foam to the affected area in response to each event. Each morning participants applied the foam they also completed the Compliance and Symptom Log, documenting the incidence and severity of night-time cramps and spasms their use of the foam and any other therapies they used to treat their night-time cramps and spasm.
- Placebo: Participants received 2, 3 ounce foam dispensers corresponding to their group (FoamA or FoamB) and a 2-week Compliance and Symptom Log. The participants were blind to the contents of the foam and the investigators until the study was completed. One foam contained Theraworx/[pH]uel (treatment) and the other contained a physiologically inert substance (placebo control).
  Placebo: Participants were instructed to apply the assigned foam to their entire upper and lower legs and feet using 8 pumps from the dispenser per leg before retiring each evening for 14 days. If participants experienced leg cramps or spasms after retiring they were instructed to reapply 2 pumps of the foam to the affected area in response to each event. Each morning participants applied the foam they also completed the Compliance and Symptom Log, documenting the incidence and severity of night-time cramps and spasms their use of the foam and any other therapies they used to treat their night-time cramps and spasm.
Period: Overall Study
Arm/Group | Theraworx | Placebo
Started | 28 | 29
Completed | 25 | 25
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Theraworx | Placebo | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Full Range); unit: years] | 47.4 [26 to 74] | 52.1 [25 to 80] | 49.8 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 39
  Male | 5 | 13 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Restless Legs Syndrome Quality of Life Instrument (RLSQoL) Over 4 Weeks
Description: Restless Legs Syndrome Quality of Life Instrument (RLSQoL) assesses the impact of restless legs symptoms on daily life, emotional well-being, social life and work life in adults 21 years and over. Each subsection is totaled separately and summed to form a total score from 0-100. Higher scores on the RLSQoL overall life impact score indicate a better quality of life. The subsections include Social Life, Daily Function, Sleep Quality, and Emotional Well-being. Each subsection questions are summed, divided by total score, and multiplied by 100 to form a scale of 0 (worst outcome) to 100 (best outcome).
Time Frame: Baseline, 2 weeks, and 4 weeks
Population: Population analyzed based off of the number of subjects who completed the study, see Overall Study Participant Flow section.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Theraworx | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale
  RLS_Social Baseline | 78.92 (4.36) | 80.75 (4.36)
  RLS_Social Week 2 | 77.75 (3.92) | 83.16 (3.92)
  RLS_Social Week 4 | 87 (3.47) | 87.03 (3.47)
  RLS_Daily Baseline | 65.33 (4.97) | 73.17 (4.97)
  RLS_Daily Week 2 | 69.50 (4.39) | 77.49 (4.39)
  RLS_Daily Week 4 | 81.50 (3.64) | 85.50 (3.64)
  RLS_Sleep Baseline | 29.56 (4.16) | 37.11 (4.16)
  RLS_Sleep Week 2 | 35.33 (3.91) | 42.04 (3.91)
  RLS_Sleep Week 4 | 47.55 (4.59) | 53.89 (4.59)
  RLS_Emotional Baseline | 58 (5.98) | 67 (5.98)
  RLS_Emotional Week 2 | 64.33 (5.51) | 72.33 (5.51)
  RLS_Emotional Week 4 | 77 (4.5) | 82.37 (4.5)
  RLS_QoL Baseline | 58.02 (4.28) | 64.51 (4.28)
  RLS_QoL Week 2 | 61.30 (3.9) | 68.29 (3.9)
  RLS_QoL Week 4 | 72.82 (3.61) | 76.29 (3.61)

2. Primary Outcome: Change in Beck Depression Scale Over 4 Weeks
Description: The Beck Depression Scale is one of the most widely used psychometric tests for measuring the severity of depression. The score is calculated by adding up the score for each of the twenty-one questions by counting the number to the right of each question marked. The highest possible total for the whole test would be sixty-three and the lowest possible score for the test would be zero. The level of depression is evaluated by: 0-10 (These ups and downs are considered normal);11-16 (Mild mood disturbance); 17-20 (Borderline clinical depression); 21-30 (Moderate depression); 31-40 (Severe depression); over 40 (Extreme depression).
Time Frame: Baseline, 2 weeks, and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Theraworx | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 12.4 (1.75) | 8.48 (1.75)
  2 Weeks | 9.56 (1.6) | 6.92 (1.6)
  4 Weeks | 6.88 (1.3) | 5.6 (1.3)

3. Primary Outcome: Change in Pittsburgh Sleep Quality Index Over 4 Weeks
Description: The Pittsburgh Sleep Quality Index is used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. The seven component scores are added together for a global score ranging from 0 to 21, 0 indicating no difficulty and 21 indicating severe difficulties.
Time Frame: Baseline, 2 weeks, and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Theraworx | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale
  Pittsburgh Sleep Quality Baseline | 10.72 (0.84) | 10.12 (0.84)
  Pittsburgh Sleep Quality Week 2 | 11 (0.83) | 9.52 (0.83)
  Pittsburgh Sleep Quality Week 4 | 9.12 (0.85) | 7.8 (0.85)

4. Primary Outcome: Change in Modified Patient Specific Functional Scale Over 4 Weeks
Description: The Modified Patient Specific Functional Scale is used to quantify activity limitation and measure functional outcome for patients with any orthopaedic condition. Three important activities that are unable to be done or are having difficulty are rated from 0 to 10, 0 being unable to perform and 10 being able to perform activity at the same level as before injury or problem. The total score is the sum of the activity scores divided by the number of activities, ranging from 0 (worst outcome) to 10 (best outcome).
Time Frame: Baseline, 2 weeks, and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Theraworx | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 4.53 (0.58) | 5.76 (0.58)
  2 Weeks | 4.99 (0.55) | 6.59 (0.55)
  4 Weeks | 6.47 (0.58) | 7.4 (0.59)

5. Secondary Outcome: Change in Symptom Log Over 4 Weeks
Description: Patients will track the number of times their leg cramps/spasms for the first 2 weeks without intervention and then how many times during the two weeks using the intervention.
Time Frame: Weeks 1, 2, 3 and 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Leg Cramps and Spasm
Arm/Group | Theraworx | Placebo
Number analyzed (Participants) | 25 | 25
Leg Cramps and Spasm
  Week 1 | 5.12 (0.34) | 4.72 (0.34)
  Week 2 | 4.72 (0.42) | 4.8 (0.42)
  Week 3 | 4.44 (0.45) | 3.32 (0.45)
  Week 4 | 3.92 (0.59) | 3.92 (0.59)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over the course of 4 weeks of participation for each subject.
Arm/Group | Theraworx | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT03159260/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03159260/Prot_SAP_001.pdf